CLINICAL TRIAL: NCT03310684
Title: The Role of the Renin-Angiotensin System in Pediatric Primary Hypertension (PHRAS)
Brief Title: Pediatric Primary Hypertension and the Renin-Angiotensin System (PHRAS)
Acronym: PHRAS
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00041266
Record Dates: First submitted 2017-10-02; First posted 2017-10-16 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-06

CONDITIONS: Pediatric Disorder; Pediatric Obesity; Primary Hypertension
Keywords: Renin-Angiotensin system; Hypertension; Obesity; Angiotensin-(1-7); Angiotensin II; FGF23; Klotho; Uric acid; Left ventricular hypertrophy
MeSH Terms: conditions — Pediatric Obesity; Essential Hypertension; Hypertension; Obesity; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypertensive: Clinical data will be collected from the electronic medical record, including height, weight, age, sex, parent-reported race, and past medical and family histories. Antihypertensive medication type and dosage will be recorded. Blood and urine samples will be collected at baseline and yearly for three years. All subjects will receive baseline and yearly echocardiograms. Subjects with overweight/obesity (BMI >=85th percentile for age and sex) will receive baseline and yearly ultrasounds of the liver to evaluate for hepatic fat infiltration. Auscultated, continuous and ambulatory blood pressure will be measured at baseline and yearly.
- Normotensive with Obesity: Clinical data will be collected from the electronic medical record, including height, weight, age, sex, parent-reported race, and past medical and family histories. Subjects will receive a baseline ultrasound of the liver to evaluate hepatic fat infiltration as per standard of care.
  Blood and urine will be collected at baseline to measure liver function (AST, ALT) and uric acid, angiotensin ll, and angiotensin-(1-7).
- Healthy Normotensive: Clinical data will be collected from the electronic medical record, including height, weight, age, sex, parent-reported race, and past medical and family histories. Subjects will have baseline echocardiograms. Blood pressure will be measured at baseline and at one year. Continuous blood pressure and ambulatory blood pressure monitoring will be assessed at baseline. Blood and urine samples will be used to measure uric acid, FGF23, klotho, and albumin, as well as the predictors angiotensin ll and angiotensin-(1-7).

SUMMARY:
Pediatric primary hypertension is increasingly common, occurring in 5-10% of normal-weight children and up to 25% of children with obesity. It is a risk factor for adult cardiovascular and renal disease. But even during childhood, hypertension is associated with significant morbidity, including cognitive impairment and organ damage. In the heart and kidneys, this organ damage is characterized by thickened heart muscle (left ventricular hypertrophy) and spillage of protein in the urine (albuminuria). Obese children are also at risk for fatty liver disease. However, the cause of pediatric primary hypertension, the role of obesity, and the mechanisms behind heart and kidney injury are poorly understood. Due to these limitations, there are no first-line medications, and treatment is often inadequate. An altered renin-angiotensin system may cause primary hypertension and related organ damage. Evidence suggests uric acid, FGF23, klotho, and obesity play a role in renin-angiotensin system-mediated injury. An improved comprehension of the pathophysiology of pediatric primary hypertension could enhance clinical care by targeting treatment to the cause of disease and informing novel measurement of organ damage.

DETAILED DESCRIPTION:
This proposal is to begin to elucidate the origins of pediatric primary hypertension and determine how it causes cardiac and renal disease. The primary hypothesis is than an altered renin-angiotensin system leads to the development of pediatric primary hypertension-related organ damage in the heart and kidney, specifically left ventricular hypertrophy and albuminuria. It is postulated that relative increase in angiotensin (Ang) ll tone compared to Ang-(1-7) tone in the circulation and the kidney (measured in the plasma and urine, respectively) leads to disease. The secondary hypotheses are that abnormalities in renin-angiotensin system tone are related to higher uric acid and FGF23, lower klotho, and, with concurrent obesity, contribute to nonalcoholic fatty liver disease. The investigators will recruit 100 subjects aged 5-17 years who are referred for a new diagnosis of pediatric primary hypertension to the Pediatric Nephrology clinic at Brenner Children's Hospital, 50 normotensive subjects with obesity recruited from the Brenner Families-in-Training program, and 10 healthy normotensive from a general pediatrics clinic in the Wake Forest Baptist Health System.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension cohort: 5 to 17 years old with a new diagnosis of pediatric primary hypertension (systolic or diastolic blood pressure >=95th percentile for age/sex/height or >=130/80 mmHg.
* Normotensive controls with obesity: 5 to 17 years old with normal systolic and diastolic blood pressure (<90th percentile for age/sex/height or <120/80 mmHg) and BMI >=85th percentile for age/sex.
* Normotensive controls: 5 to 17 years old with normal systolic and diastolic blood pressure (<90th percentile for age/sex/height or <120/80 mmHg).

Exclusion Criteria:

* Secondary hypertension
* Confounding medical condition (e.g. diabetes mellitus, chronic kidney disease, heart disease, vascular disease, inflammatory or rheumatologic disease)
* Non-English and non-Spanish speaking
* Inability to complete assessments

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients of the Pediatric Nephrology Clinic and Pediatric Gastroenterology Clinic at Brenner Children's Hospital. Patients from a general pediatric clinic at Wake Forest Baptist Health.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Left ventricular hypertrophy | Yearly for 3 years
  Left ventricular hypertrophy according to elevated left ventricular mass index (>51 g/m^2.7 (>8 years of age, both sexes) or >115 g/body surface area (males) and >95 g/body surface area (females)) on serial echocardiogram.

SECONDARY OUTCOMES:
Albuminuria | Yearly for 3 years
  Albumin-to-creatinine ratio >30 mg/g
Ambulatory systolic blood pressure load | Yearly for 3 years
  Percent of 24-hour ambulatory systolic blood pressure above the 95th percentile (>25% abnormal)
Ambulatory diastolic blood pressure load | Yearly for 3 years
  Percent of 24-hour ambulatory diastolic blood pressure above the 95th percentile (>25% abnormal)
Ambulatory systolic blood pressure nocturnal dipping | Yearly for 3 years
  Percent of 24-hour ambulatory systolic blood pressure that drops below the mean blood pressure overnight
Ambulatory diastolic blood pressure nocturnal dipping | Yearly for 3 years
  Percent of 24-hour ambulatory diastolic blood pressure that drops below the mean blood pressure overnight
Clinic systolic blood pressure | Yearly for 3 years
  Auscultated systolic blood pressure (mmHg)
Clinic diastolic blood pressure | Yearly for 3 years
  Auscultated diastolic blood pressure (mmHg)
Nonalcoholic fatty liver disease | Yearly for 3 years
  Fat infiltration (yes or no) as measured on liver ultrasound with elastography in subjects with overweight/obesity (BMI >=85th percentile)
Continuous systolic blood pressure | Yearly for 3 years
  Systolic blood pressure measured continuously for 10 minutes (mmHg)
Continuous diastolic blood pressure | Yearly for 3 years
  Diastolic blood pressure measured continuously for 10 minutes (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M South, MD MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Din-Dzietham R, Liu Y, Bielo MV, Shamsa F. High blood pressure trends in children and adolescents in national surveys, 1963 to 2002. Circulation. 2007 Sep 25;116(13):1488-96. doi: 10.1161/CIRCULATIONAHA.106.683243. Epub 2007 Sep 10. PMID 17846287
- [Background] Richey PA, Disessa TG, Somes GW, Alpert BS, Jones DP. Left ventricular geometry in children and adolescents with primary hypertension. Am J Hypertens. 2010 Jan;23(1):24-9. doi: 10.1038/ajh.2009.164. Epub 2009 Oct 22. PMID 19851297
- [Background] Iyer SN, Ferrario CM, Chappell MC. Angiotensin-(1-7) contributes to the antihypertensive effects of blockade of the renin-angiotensin system. Hypertension. 1998 Jan;31(1 Pt 2):356-61. doi: 10.1161/01.hyp.31.1.356. PMID 9453328
- [Background] Shaltout HA, Rose JC, Chappell MC, Diz DI. Angiotensin-(1-7) deficiency and baroreflex impairment precede the antenatal Betamethasone exposure-induced elevation in blood pressure. Hypertension. 2012 Feb;59(2):453-8. doi: 10.1161/HYPERTENSIONAHA.111.185876. Epub 2012 Jan 3. PMID 22215705
- [Background] Simoes E Silva AC, Diniz JS, Regueira Filho A, Santos RA. The renin angiotensin system in childhood hypertension: selective increase of angiotensin-(1-7) in essential hypertension. J Pediatr. 2004 Jul;145(1):93-8. doi: 10.1016/j.jpeds.2004.03.055. PMID 15238914
- [Background] South AM, Nixon PA, Chappell MC, Diz DI, Russell GB, Snively BM, Shaltout HA, Rose JC, O'Shea TM, Washburn LK. Antenatal corticosteroids and the renin-angiotensin-aldosterone system in adolescents born preterm. Pediatr Res. 2017 Jan;81(1-1):88-93. doi: 10.1038/pr.2016.179. Epub 2016 Sep 16. PMID 27636897
- [Background] Ferrario CM, Martell N, Yunis C, Flack JM, Chappell MC, Brosnihan KB, Dean RH, Fernandez A, Novikov SV, Pinillas C, Luque M. Characterization of angiotensin-(1-7) in the urine of normal and essential hypertensive subjects. Am J Hypertens. 1998 Feb;11(2):137-46. doi: 10.1016/s0895-7061(97)00400-7. PMID 9524041
- [Background] Washburn LK, Nixon PA, Russell GB, Snively BM, O'Shea TM. Preterm Birth Is Associated with Higher Uric Acid Levels in Adolescents. J Pediatr. 2015 Jul;167(1):76-80. doi: 10.1016/j.jpeds.2015.03.043. Epub 2015 Apr 11. PMID 25868431
- [Background] Feig DI, Soletsky B, Johnson RJ. Effect of allopurinol on blood pressure of adolescents with newly diagnosed essential hypertension: a randomized trial. JAMA. 2008 Aug 27;300(8):924-32. doi: 10.1001/jama.300.8.924. PMID 18728266
- [Background] Mazzali M, Hughes J, Kim YG, Jefferson JA, Kang DH, Gordon KL, Lan HY, Kivlighn S, Johnson RJ. Elevated uric acid increases blood pressure in the rat by a novel crystal-independent mechanism. Hypertension. 2001 Nov;38(5):1101-6. doi: 10.1161/hy1101.092839. PMID 11711505
- [Background] Seeherunvong W, Abitbol CL, Chandar J, Rusconi P, Zilleruelo GE, Freundlich M. Fibroblast growth factor 23 and left ventricular hypertrophy in children on dialysis. Pediatr Nephrol. 2012 Nov;27(11):2129-2136. doi: 10.1007/s00467-012-2224-7. Epub 2012 Jun 19. PMID 22710695
- [Background] Engeli S, Bohnke J, Gorzelniak K, Janke J, Schling P, Bader M, Luft FC, Sharma AM. Weight loss and the renin-angiotensin-aldosterone system. Hypertension. 2005 Mar;45(3):356-62. doi: 10.1161/01.HYP.0000154361.47683.d3. Epub 2005 Jan 3. PMID 15630041
- [Background] Zhang H, Yang H, Lai C, Xu X, Huang K, Fu J. Quantitative relationship between liver fat content and metabolic syndrome in obese children and adolescents. Clin Endocrinol (Oxf). 2015 Jul;83(1):43-9. doi: 10.1111/cen.12758. Epub 2015 Mar 16. PMID 25711346
- [Background] Kuczmarski RJ, Ogden CL, Guo SS, Grummer-Strawn LM, Flegal KM, Mei Z, Wei R, Curtin LR, Roche AF, Johnson CL. 2000 CDC Growth Charts for the United States: methods and development. Vital Health Stat 11. 2002 May;(246):1-190. PMID 12043359
- [Background] Schwartz GJ, Brion LP, Spitzer A. The use of plasma creatinine concentration for estimating glomerular filtration rate in infants, children, and adolescents. Pediatr Clin North Am. 1987 Jun;34(3):571-90. doi: 10.1016/s0031-3955(16)36251-4. PMID 3588043
- [Background] Fortunato JE, Tegeler CL, Gerdes L, Lee SW, Pajewski NM, Franco ME, Cook JF, Shaltout HA, Tegeler CH. Use of an allostatic neurotechnology by adolescents with postural orthostatic tachycardia syndrome (POTS) is associated with improvements in heart rate variability and changes in temporal lobe electrical activity. Exp Brain Res. 2016 Mar;234(3):791-8. doi: 10.1007/s00221-015-4499-y. Epub 2015 Dec 8. PMID 26645307
- [Background] Flynn JT, Daniels SR, Hayman LL, Maahs DM, McCrindle BW, Mitsnefes M, Zachariah JP, Urbina EM; American Heart Association Atherosclerosis, Hypertension and Obesity in Youth Committee of the Council on Cardiovascular Disease in the Young. Update: ambulatory blood pressure monitoring in children and adolescents: a scientific statement from the American Heart Association. Hypertension. 2014 May;63(5):1116-35. doi: 10.1161/HYP.0000000000000007. Epub 2014 Mar 3. No abstract available. PMID 24591341
- [Background] Khoury PR, Mitsnefes M, Daniels SR, Kimball TR. Age-specific reference intervals for indexed left ventricular mass in children. J Am Soc Echocardiogr. 2009 Jun;22(6):709-14. doi: 10.1016/j.echo.2009.03.003. Epub 2009 May 7. PMID 19423289
- [Background] Rademacher ER, Sinaiko AR. Albuminuria in children. Curr Opin Nephrol Hypertens. 2009 May;18(3):246-51. doi: 10.1097/MNH.0b013e3283294b98. PMID 19276802
- [Background] Assadi F. Effect of microalbuminuria lowering on regression of left ventricular hypertrophy in children and adolescents with essential hypertension. Pediatr Cardiol. 2007 Jan-Feb;28(1):27-33. doi: 10.1007/s00246-006-1390-4. Epub 2007 Feb 16. PMID 17308944

DOCUMENTS (2):
  • Study Protocol (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03310684/Prot_000.pdf
  • Informed Consent Form (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT03310684/ICF_001.pdf